CLINICAL TRIAL: NCT03684278
Title: Phase IIb, Randomised, Double-blind, Placebo-controlled, Multi-centre Trial of Infliximab With Transcriptomic Biomarker and Mechanism Evaluation in Patients With Acute Pancreatitis.
Brief Title: Randomised Treatment of Acute Pancreatitis With Infliximab: Double-blind, Placebo-controlled, Multi-centre Trial (RAPID-I)
Acronym: RAPID-I
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Bangor University (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); Medical Research Council (Other Government); National Institute for Health Research, United Kingdom (Other Government); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UoL001326; 2017-003840-19 (EudraCT Number); 15/20/01 (Other Grant/Funding Number: MRC and NIHR EME)
Record Dates: First submitted 2018-07-04; First posted 2018-09-25 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Infliximab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: RAPID-I is a randomised, placebo-controlled, double-blind, multi-centre, three-arm, phase IIb efficacy trial of infliximab in patients with AP. Patients will be randomised (1:1:1 allocation ratio) to receive an intravenous infusion of either 5 mg/kg or 10 mg/kg infliximab or placebo, initiated within 36 hours of admission to hospital with acute pancreatitis. Treatment allocation will only be revealed to those responsible for trial treatment preparation (Pharmacy or an independent research team not administering the trial medication) to ensure the research team administering the treatment remains blinded.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Once the delegated research team member performs randomisation and the staff member responsible for preparation of trial medication is provided with the allocation to either Arm A, B or C, that latter staff member will prepare the infusion, which will be covered by an opaque sleeve and labelled for blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Infusion of 5 mg/kg Infliximab (Active Comparator): Infliximab (Remicade) to be administered as a one time intravenous infusion in 250 ml (500 ml if patient weighs over 100 kg) 0.9% sodium chloride solution over a period of 2 hours. Dosage calculated at 5 mg of Infliximab, per kg of patient body weight.
  Interventions: Drug: Infusion of 5 mg/kg Infliximab
- Infusion of 10 mg/kg Infliximab (Active Comparator): Infliximab (Remicade) to be administered as a one time intravenous infusion in 250 ml (500 ml if patient weighs over 100 kg) 0.9% sodium chloride solution over a period of 2 hours. Dosage calculated at 10 mg of Infliximab, per kg of patient body weight.
  Interventions: Drug: Infusion of 10 mg/kg Infliximab
- 0.9% Sodium Chloride (Placebo) (Placebo Comparator): 250 ml (500 ml if patient weighs over 100 kg) 0.9% Sodium Chloride to be administered as a one time intravenous infusion over a period of 2 hours.
  Interventions: Other: 0.9% Sodium Chloride (Placebo)

INTERVENTIONS:
Drug: Infusion of 5 mg/kg Infliximab — Infliximab is a prescription drug with marketing authorisation for the treatment of rheumatoid arthritis, Crohn's disease, ulcerative colitis, ankylosing spondylitis, psoriatic arthritis and psoriasis. In the RAPID-I trial infliximab will be used outside the manufacturer's indication for the treatment of AP, and it is classed as an investigational medicinal product (IMP).
  Other Names: Remicade
  Arms: Infusion of 5 mg/kg Infliximab
Drug: Infusion of 10 mg/kg Infliximab — Infliximab is a prescription drug with marketing authorisation for the treatment of rheumatoid arthritis, Crohn's disease, ulcerative colitis, ankylosing spondylitis, psoriatic arthritis and psoriasis. In the RAPID-I trial infliximab will be used outside the manufacturer's indication for the treatment of AP, and it is classed as an investigational medicinal product (IMP).
  Other Names: Remicade
  Arms: Infusion of 10 mg/kg Infliximab
Other: 0.9% Sodium Chloride (Placebo) — 250 ml (500 ml if patient weighs over 100 kg) of 0.9% Sodium Chloride
  Arms: 0.9% Sodium Chloride (Placebo)

SUMMARY:
This study evaluates the effectiveness and safety of infliximab in the treatment of acute pancreatitis in adults. A third of participants will receive one single dose of infliximab via infusion, another third will receive a higher dose of infliximab via infusion and the final third of participants will receive a placebo infusion.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is an inflammatory disorder of the pancreas causing excruciating pain, gastrointestinal dysfunction and pronounced systemic inflammatory responses with circulatory and respiratory disturbances that can lead to organ failure and death.

Tumour necrosis factor alpha (TNFα) has a major role in the pathogenesis and severity of acute pancreatitis. TNFα levels rise early and remain elevated for days in human AP, proportional to severity, presenting a suitable drug target to inhibit the amplified immune responses that further damage the pancreas and drive widespread organ dysfunction.

Infliximab is a chimeric monoclonal antibody biologic drug that blocks the actions of tumor necrosis factor alpha (TNF-α) and is normally used to treat autoimmune diseases. Infliximab has been selected as it is given via intravenous infusion, which will ensure rapid bioavailability to treat AP. This is different from most other biologics, which are given subcutaneously.

This trial will determine the efficacy of early initiation of anti-TNF treatment in AP, setting new standards for trials in AP. Using a randomised, double-blind, placebo-controlled adaptive design, with two doses of a single intravenous infusion of infliximab at 5 mg/kg or 10 mg/kg, the trial will determine size of any effect and safety of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients attending Accident and Emergency (A&E) at or admitted to recruiting hospitals via a GP with a new diagnosis of AP established by two of the following three criteria: (1) typical continuous upper abdominal pain; (2) amylase and/or lipase three or more times the upper limit of normal; (3) characteristic findings on abdominal imaging (if undertaken urgently by CT or MRI)
* Patients in whom trial treatment can be started within 36 hours of admission to hospital with a new diagnosis of acute pancreatitis allowing 120 min for preparation of trial medication
* Patients from whom appropriate consent is obtained (from the patient or their legal representative).

Exclusion Criteria:

* Age <18 or >85
* Patients with a bodyweight over 200 kg
* Known previous AP within the last 30 days or chronic pancreatitis
* Multiple sclerosis, systemic vasculitis, Guillain-Barré syndrome or other demyelinating disorder
* Known epilepsy
* Moderate to severe heart failure and/or coronary disease (NYHA III/IV)
* Severe respiratory conditions including cystic fibrosis, severe asthma and severe chronic obstructive pulmonary disease (COPD)
* On home oxygen or home mechanical ventilation
* Jaundice and/or known advanced liver disease
* Known cancer for which chemotherapy and/or radiotherapy ongoing/completed in last 6 months
* Known haematological malignancy
* Known cancer with palliative care
* Known established infection prior to or suspected infection, including COVID-19, at the time of AP onset
* Known history of tuberculosis, or household contact with those with tuberculosis or opportunistic infection
* Known history of infective hepatitis
* Rare diseases or inborn errors of metabolism that significantly increase the risk of infections, including severe combined immunodeficiency (SCID) and homozygous sickle cell disease
* Known live vaccine or infectious agent within one month of admission
* Known immunosuppressive or biologic therapy within one month of admission
* Known hypersensitivity to infliximab or to inactive components of REMICADE® or to any murine proteins
* Known pregnancy or lactation at admission
* Females of childbearing potential who do not agree to use adequate contraception up to 6 months after infliximab infusion
* Known participation in investigational medicinal product study within last three months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Difference in mean serum CRP measured on days 2, 4 and 14 | Days 2, 4 (+/- 1 day), and 14 (+/- 2 days)
  Difference in mean serum CRP measured on (summated as AUC) in the active arms (5 mg/kg or 10 mg/kg) versus the placebo arm. CRP assays will be undertaken on blood samples centrally to ensure standardised measurement, and when central measurements of CRP at specific time points are not available for any patient, CRP measures from that patient's specific recruiting centre will be sought.

SECONDARY OUTCOMES:
Pain scores | First 14 Days
  Patient will complete a Numerical Rating Scale.The scale is from 0-10 (0= no pain and 10 = worst pain possible)
Opiate requirements | First 14 days
  Recording of daily morphine equivalents by research team
Nutritional deficit | First 14 days
  Number of days without solid food for first 14 days
Decline in serum albumen | First 14 days
  Albumen measured via blood samples
Rise in neutrophils | First 14 days
  Neutrophils measured in blood samples
Sequential organ failure assessment (SOFA) score | First 14 days
  Summed respiratory (0-4), cardiovascular (0-4) and renal (0-4) SOFA scores on each of the first 28 days after hospital admission
Local pancreatic injury | Day 14 +/- 7 days
  Contrast-enhanced CT scan assessed by a central panel
Revised Atlanta Classification (RAC) | 90 days after admission
  RAC severity classification (mild, moderate or severe)
Infective complications | First 90 days
  Infective complications reported
Length of hospital stay | Up to 90 days
  Length of time patient remains within hospital as an inpatient
Mortality | Within the first 90 days
  Patient death
Patient reported outcome | Day 4, Day 14 and Day 90
  EuroQol EQ-5D-5L
Potential safety signals | Up to 90 days
  Adverse events relating to infliximab including infusion reactions and delayed serum sickness reactions
Anti-infliximab antibody concentration | Day 14
  Blood sample analysis to determine the concentration of anti-infliximab antibodies
Incremental cost per quality adjusted life years (QALY) gained by trial treatment | Days 4, 14 and 90
  QALYs using data from the EQ-5D-5L questionnaire
Infliximab concentration | Day 14
  Infliximab measured in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sutton, DPhil, FRCS, Principal Investigator — University of Liverpool
Locations (13):
- United Kingdom (13):
  - Aberdeen Royal Infirmary, Aberdeen, Aberdeenshire
  - University Hospital of Wales, Cardiff, Cardiff
  - Royal Cornwall Hospital, Truro, Cornwall
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - University College London Hospital, London, Greater London
  - St Mary's Hospital, London, Greater London
  - Charing Cross Hospital, London, Greater London
  - Royal Liverpool University Hospital, Liverpool, Merseyside
  - Aintree University Hospital, Liverpool, Merseyside
  - Whiston Hospital, Whiston, Merseyside
  - Queen's Medical Centre, Nottingham, Nottinghamshire
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - St James's University Hospital, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: No